CLINICAL TRIAL: NCT05855356
Title: The Long-CoviD Patients Causal Diagnosis and Rehabilitation Randomized Feasibility Controlled Trial in Patients With Dysautonomia: the LoCoDiRe-Dys Study
Brief Title: Post Covid-19 Dysautonomia Rehabilitation Randomized Controlled Trial
Acronym: LoCoDiRe-Dys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evangelismos Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other); LONG COVID GREECE (Unknown); 414 Military Hospital of Special Diseases (Unknown)
Responsible Party: Principal Investigator, Antonios Kontaxakis, PM&R Consultant, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22
Record Dates: First submitted 2023-05-08; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Post-Acute COVID-19 Syndrome; Dysautonomia
Keywords: Long Covid; Post Covid-19 condition; Rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Autonomic Nervous System Diseases | interventions — Rehabilitation; Standard of Care

STUDY DESIGN:
Intervention Model Description: unblinded randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LoCoDiRe-Dys (Experimental): Respiratory physiotherapy, personalized aerobic and strength training in parallel with standard of care
  Interventions: Procedure: Rehabilitation; Procedure: Standard of Care
- Standard of Care (Active Comparator): Standard of care including behavioural and medical advice
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: Rehabilitation — respiratory physiotherapy, personalized aerobic and strength training
  Arms: LoCoDiRe-Dys
Procedure: Standard of Care — Behavioural and Medical management

SUMMARY:
Dysautonomia in post-covid-19 condition appears to affect a significant number of patients, with reports raising the incidence up to 61%, having an overlap with myalgic encephalomyelitis/ chronic fatigue syndrome. Quality of life and daily function is significantly impacted and conservative management interventions, despite the lack of high quality evidence up to now, are needed to ameliorate disability. 50 adults with a dysautonomia post-covid-19 diagnosis based on the Ewing battery and a NASA lean test will be enrolled in a randomized single blinded controlled trial with a crossover design. Feasibility and lack of definite dysautonomia diagnosis will be the primary out-comes, while secondary outcomes will be health-related, clinical and cardiopulmonary exercise test indicators. Safety and acceptance will also be checked, primarily excluding participants with post exertional malaise. The Long-CoViD patients Causal Diagnosis and Rehabilitation study in patients with Dysautonomia (LoCoDiRE-Dys) study intervention will consist of an educational module, breathing retraining and an individualized exercise intervention of biweekly sessions for two months with regular assessment of both groups. LoCoDiRe- Dys aims to be the first post-covid-19 randomized study in people with dysautonomia offering a multimodal intervention both in diagnosis and management

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* WHO definition of post covid-19 condition
* Confirmed dysautonomia diagnosis through Ewing Battery
* Able to attend 2 times/ week for 8 weeks
* Able to provide informed consent

Exclusion Criteria:

* Absolute or relative contra-indications to exercise due to cardiac pathology
* Serious mental/ cognitive impairment that will not allow systematic participation
* Unable to regularly reach the center
* Pregnancy
* CFS/ME fulfilling the Canadian Consensus Criteria
* Secondary health conditions that would explain symptoms, intervene in dysautonomia diagnosis or would impede participation in the exercise protocol (i.e. , untreated hypothyroidism and Diabetes Melitus, major psychiatric disorders, COPD, PICS, Pulmonary Fibrosis, chronic respiratory or heart failure, not ambulatory, suffering from dementia, chronically paralyzed, with paraplegia, with multiple injuries or other serious orthopedic problems that caused disability, patients suffering from very serious underlying diseases such as end-stage cancer, and those with neurological diseases causing disability)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Number of patients with lack of definite Dysautonomia Diagnosis | 4 months
  Ewing Battery is a validated instrument to diagnose dysautonomia, with a definite diagnosis when 2 out of 4 heart rate tests are abnormal
Compliance, Adverse Events and Protocol Titration to examine feasibility of the trial | 4 months
  Process measures that will substantiate offering of the service

SECONDARY OUTCOMES:
10 minutes NASA Lean Test | checked at [0], [8] and [16] weeks
  Validated measure to record orthostatic intolerance, recording of blood pressure and heart rate in 5 min supine position, and every minute when standing up till 10 min
Six minute Walk Test | checked at [0], [8] and [16] weeks
  Validated measure, a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
1 minute sit to stand test | checked at [0], [8] and [16] weeks
  Validated measure to record the times standing up from a chair, closely related with cardiorespiratory capacity and lower limb strength
Fatigue Severity Scale | checked at [0], [8] and [16] weeks
  Validated measure to record fatigue severity as reported by the patient, 9 statements each in a scale of 1-7, min 9 max 63
modified Medical Research Council Dyspnea Scale | checked at [0], [8] and [16] weeks
  Validated measure to record functional disability because of dyspnea as reported by the patient in a scale 0-4
Nijmegen Questionnaire | checked at [0], [8] and [16] weeks
  Validated measure to record dysfunctional breathing as recorded by the patient with each statement valued 0-4, with A score of over 23 out of 64 suggest a positive diagnosis of hyperventilation syndrome.
Montreal Cognitive Assessment | checked at [0], [8] and [16] weeks
  Validated measure for rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation, with a normal score over 25/30
International Physical Activity Questionnaire | checked at [0], [8] and [16] weeks
  Validated measure with 27 item self reporting physical activity of the patient
Hospital Anxiety and Depression Scale | checked at [0], [8] and [16] weeks
  Validated measure, a 14-item measure designed to assess anxiety and depression symptoms in medical patients. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case
EuroQoL 5 Dimensions 5 Levels | checked at [0], [8] and [16] weeks
  Validated measure, a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Cardiorespiratory exercise test | checked at [0], [8] and [16] weeks
  A specialized type of stress test or exercise test that measures exercise ability
Lower Extremity Strength | checked at [0], [8] and [16] weeks
  Assessment of lower extremity strength using a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Katsaounou, Study Director — Director of the Lond Covid Outpatient Clinic
Locations (1):
- First Department of Critical Care Medicine and Pulmonary Services, Evangelismos Hospital, National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Anonymized clinical data
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 3 months after completion of the study, for 5 years on
Access Criteria: Request reasons clearly stated- Sharing of further analysis plan

REFERENCES:
- [Background] Ormiston CK, Swiatkiewicz I, Taub PR. Postural orthostatic tachycardia syndrome as a sequela of COVID-19. Heart Rhythm. 2022 Nov;19(11):1880-1889. doi: 10.1016/j.hrthm.2022.07.014. Epub 2022 Jul 16. PMID 35853576
- [Background] Raj SR, Guzman JC, Harvey P, Richer L, Schondorf R, Seifer C, Thibodeau-Jarry N, Sheldon RS. Canadian Cardiovascular Society Position Statement on Postural Orthostatic Tachycardia Syndrome (POTS) and Related Disorders of Chronic Orthostatic Intolerance. Can J Cardiol. 2020 Mar;36(3):357-372. doi: 10.1016/j.cjca.2019.12.024. PMID 32145864
- [Background] Katsarou MS, Iasonidou E, Osarogue A, Kalafatis E, Stefanatou M, Pappa S, Gatzonis S, Verentzioti A, Gounopoulos P, Demponeras C, Konstantinidou E, Drakoulis N, Asimakos A, Antonoglou A, Mavronasou A, Spetsioti S, Kotanidou A, Katsaounou P. The Greek Collaborative Long COVID Study: Non-Hospitalized and Hospitalized Patients Share Similar Symptom Patterns. J Pers Med. 2022 Jun 17;12(6):987. doi: 10.3390/jpm12060987. PMID 35743774